CLINICAL TRIAL: NCT07274813
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of HLX37 (Recombinant Human Bispecific Antibodies Against PD-L1 and VEGF) in Patients With Advanced/Metastatic Solid Tumors
Brief Title: A Phase I Study to Evaluate the Safety, Tolerability, and PK of HLX37 in Advanced/Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HLX37- FIH101
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Advanced/Metastatic Solid Tumors; NSCLC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ia (Dose Escalation) (Experimental): Patients with advanced/metastatic solid tumors
  Interventions: Drug: HLX37-Dose1; Drug: HLX37-Dose2; Drug: HLX37-Dose3; Drug: HLX37-Dose4

INTERVENTIONS:
Drug: HLX37-Dose1 — Patients with advanced/metastatic solid tumors
Drug: HLX37-Dose2 — 5mg/kg Q3W
Drug: HLX37-Dose3 — 10mg/kg Q3W
Drug: HLX37-Dose4 — 20mg/kg Q3W

SUMMARY:
This study is an open-label first-in-human phase I clinical study to evaluate the safety, tolerability, and pharmacokinetic characteristics of HLX37 in patients with advanced/metastatic solid tumors.

DETAILED DESCRIPTION:
This study is an open-label first-in-human phase I clinical study to evaluate the safety, tolerability , and pharmacokinetic characteristics of HLX37 with escalated doses in the treatment of patients with advanced/metastatic solid tumors.

In Phase Ia Part 1of this study, a 3 + 3 dose escalation method will be adopted, and the patients will be administered with HLX37 at different doses via intravenous infusion. The DLT observation period lasts for 3 weeks after the first administration of HLX37.

After the DLT observation period of the single-drug ramp-up 20mg/kg dose group ended and the SRC safety assessment was conducted, that is Initiate the Phase Ia Part2 of this study to conduct HLX37 in patients with advanced non-small cell lung cancerThe dosage of combined chemotherapy is increasing. The 3+3 dose escalation method will be adopted, and the subjects will receive different doses. Intravenous infusion administration of HLX37 in combination with chemotherapy (tentatively 10 mg/kg, 20 mg/kg, 30 mg/kg) Or other doses of HLX37 combined with chemotherapy, administered intravenously at Q3W. DLT observation period 3 weeks after the first administration of HLX37 in combination with chemotherapy.

In phase Ib of this study, The Safety Review Committee will recommend dose groups for expansion based on the safety, efficacy and PK data of the dose escalation phase.

ELIGIBILITY:
Selection criteria Before the trial, fully understand the content, process and possible adverse reactions of the trial, sign the informed consent form, voluntarily participate in the trial, and be able to complete the research in accordance with the requirements of the trial protocol.

2. At the time of signing the ICF, the applicant must be at least 18 years old and no more than 75 years old, with no gender restrictions.

3. part 1 of Stage Ia enrolled subjects with advanced or metastatic solid tumors confirmed by histology or cytology, who had failed at least one standard systemic treatment in the advanced or metastatic stage of the disease (subjects who had received neoadjuvant or adjuvant therapy, if disease progression or recurrence occurred within 6 months after the end of treatment) Then this treatment plan will be regarded as a failure of standard treatment, or there is currently no effective standard treatment method.

Part 2 of stage Ia enrollment confirmed by histology or cytology Locally advanced (stage ⅢB/ⅢC) or metastatic (stage IV) NSCLC that is not suitable for radical treatment (complete surgical resection, concurrent/sequential chemoradiotherapy) (according to the 8th edition of lung cancer TNM staging by the Union for International Cancer Control and the American Joint Committee on Cancer AJCC), and should meet the following criteria:

Subjects without targeted driver gene alterations (AGA) :

For non-squamous NSCLC subjects, there must be previous test results confirming negative EGFR and ALK gene alterations. If there are no previous EGFR and ALK test results, the subjects are required to undergo relevant tests at the research center. For subjects with squamous NSCLC, if the previous EGFR and/or ALK gene status is unknown, corresponding tests are not required before enrollment in this study.

There are no known alterations in the targeted driver genes of ROS1, NTRK, BRAF, METexon 14 skipping or RET.

· Has not received systematic anti-tumor treatment 2) Subjects with AGA: There must be previous test results confirming the existence of one or more targeted driver gene alterations.

Previous failure of at least one line of standard treatment should include at least targeted therapy for driver gene alterations (patients with EGFR mutations must be treated with EGFR inhibitors).

For stage Ib, sensitive advanced solid tumor types will be selected for exploration based on the results of stage Ia.

4. Within 4 weeks before the first administration, at least one measurable lesion was present according to the efficacy evaluation criteria of RECIST 1.1. For patients who have received radiotherapy before, if the lesion can be measured according to RECIST v1.1 and there is objective evidence proving significant progression after radiotherapy, the lesion that has undergone radiotherapy can be regarded as the target lesion. Brain metastases cannot be used as target lesions.

5. Seven days before the first administration, the ECOG physical strength score is 0-1.

6. The expected survival period exceeds 3 months; 7. Before the first study of drug administration, there must be an interval of at least 28 days from previous major surgical operations, medical device treatment, local radiotherapy (except palliative radiotherapy for bone lesions), cytotoxic chemotherapy, immunotherapy or biologics treatment. There should be at least a 14-day interval from previous small molecule targeted drug therapy and hormone therapy. There should be at least a 7-day interval from traditional Chinese medicine treatment or minor surgery with anti-tumor indications. And the AE caused by the treatment recovered to CTCAE v5.0 ≤ grade 1 (excluding alopecia); 8. The subject agrees to provide archived tumor tissue specimens that meet the testing requirements (from the most recent surgery or biopsy, preferably within 2 years) or agrees to undergo biopsy to collect tumor tissue for PD-L1 expression testing; Note: The subjects are required to provide tumor samples (paraffin blocks or unstained sections, which must meet the quality control standards for testing) collected from non-radiotherapy sites during or after the diagnosis of malignant tumors and treated with formalin-fixed paraffin embedding (FFPE), as well as the relevant pathological reports of the above specimens.

9. Laboratory tests within 7 days before the first administration of the study confirmed adequate organ function (no blood transfusion or granulocyte colony-stimulating factor was received within 14 days before the first administration) : 10.The Child-Pugh score of the subjects with hepatocellular carcinoma must be A.

11.Male and female subjects of fertility must agree to use at least one highly effective contraceptive method for contraception during the trial and for at least six months after the last administration of the study drug. Female subjects of childbearing age must have a negative pregnancy test result within 7 days prior to enrollment.

Exclusion criteria

Subjects who meet any of the following criteria will not be eligible for this study:

1. There should be a history of other malignant tumors within 3 years prior to the first medication, except for cured cervical carcinoma in situ or basal cell carcinoma of the skin.
2. There have been adverse events in the past that led to the permanent termination of immunotherapy; Or there was a history of grade ≥2 immune-related pneumonia or immune-related myocarditis;
3. Has a history of (non-infectious) interstitial lung disease (ILD), and currently still requires steroid drug treatment; Or currently having active ILD, or suspected through imaging researchers at the time of screening that there is a risk of ILD aggravation or that they are not suitable to participate in this study;
4. It is known that the subject has had a severe allergic reaction to macromolecular protein preparations/monoclonal antibodies in the past, or is allergic to the components of the test drug preparation;
5. Within two weeks before the first medication, there is an active systemic infectious disease that requires intravenous antibiotic treatment;
6. The subjects have poorly controlled clinical symptoms or diseases of the cardiovascular and cerebrovascular system, including but not limited to: (1) NYHA grade II or above heart failure or left ventricular ejection fraction (LVEF) < 50%; (2) Unstable angina pectoris; (3) Has experienced myocardial infarction or cerebrovascular accident within 6 months (excluding lacunar infarction, mild cerebral ischemia or transient ischemic attack); (4) Poorly controlled arrhythmias (including QTc intervals of ≥ 450 ms in men and ≥ 470 ms in women) (QTc intervals are calculated using the Fridericia formula);
7. Subjects who had experienced the following diseases within 12 months prior to the first administration: a history of lower esophageal varices, severe ulcers, unhealed wounds, gastrointestinal perforation, abdominal fistula, gastrointestinal obstruction, abdominal abscess or a history of acute gastrointestinal bleeding; Subjects who have experienced the following diseases within 6 months prior to the first administration: any arterial thromboembolic event, NCI CTCAE V.5.0 grade 3 or higher venous thromboembolism, transient ischemic attack, cerebrovascular accident, hypertensive crisis or history of hypertensive encephalopathy, subjects with history of acute exacerbation of chronic obstructive pulmonary disease; Patients currently suffering from hypertension with a systolic blood pressure of ≥160 MMHG or a diastolic blood pressure of ≥100 MMHG after oral antihypertensive drug treatment.
8. Known to have meningeal metastasis, or uncontrolled or symptomatic central nervous system (CNS) metastasis, manifested as clinical symptoms, cerebral edema, spinal cord compression and/or progressive growth. Subjects with a history of central nervous system metastasis or spinal cord compression who have clearly received treatment and have been determined by the investigator to have stable clinical manifestations after discontinuing anticonvulsants and steroids for 8 weeks before the start of the study treatment can be enrolled in the study. Untreated, asymptomatic subjects with brain metastases (i.e., those without neurological symptoms, no need for corticosteroid hormones, no long diameter of any brain metastases >1.5 cm, and no obvious edema around the brain metastases) can be enrolled. Brain metastases are not regarded as target lesions.
9. There is a known active or suspected autoimmune disease. However, subjects with autoimmune hypothyroidism who have received thyroid hormone replacement therapy are allowed to participate in the study; Allow controlled type 1 diabetes subjects receiving insulin treatment to participate in the study;

Subjects who have received systemic corticosteroids (prednisone > 10mg/ day or equivalent doses of similar drugs) or other immunosuppressants within 14 days prior to the first administration; Except for the following situations: treatment with topical, ocular, intra-articular, intranasal and inhaled corticosteroids; Short-term use of corticosteroids for preventive treatment in cases such as contrast agents;

11. Suffering from active pulmonary tuberculosis;

12. Subjects with a history of severe bleeding tendencies or coagulation disorders; Subjects with clinically significant bleeding symptoms within one month before the first administration, including but not limited to gastrointestinal bleeding, hemoptysis (defined as coughing up or expelling ≥1 teaspoon of fresh blood or small blood clots, or only coughing up blood without sputum; those with sputum blood can be included), and epistaxis (excluding epistaxis and bloody reflux mucus); Subjects whose imaging examinations during screening showed that the tumor surrounded important blood vessels or had obvious necrosis and cavities, and the researchers judged that there was a risk of bleeding in participating in the study; Patients with central and cavitary squamous non-small cell lung cancer (according to the researchers' judgment, such patients have a higher risk of bleeding).

13. Currently using or having used aspirin (> 325mg/ day) or dipyridamole, clopidine, clopidogrel and cilostazole for treatment within 7 days before the first use.

14. Currently in use or under study, full-dose oral or injectable anticoagulant drugs or thrombolytic drugs have been used for therapeutic purposes within 7 days prior to the first administration. Prophylactic anticoagulant therapy is permitted for open intravenous infusion systems, provided that the drug activity is less than 1.5 times the upper limit of normal for the international normalized ratio (INR) and the partial thromboplastin time (APTT) is within the normal range within 14 days prior to the first administration. Prophylactic use of low-molecular-weight heparin (i.e. Enoxaparin 40mg/ day) is permitted.

15. Daily administration of non-steroidal anti-inflammatory drugs is required for long-term treatment. Occasional use of NSAIDs is permitted to relieve medical symptoms such as headache or fever 16. In the past, when receiving anti-angiogenic therapy, grade ≥3 toxicity related to anti-angiogenic therapy occurred (except for toxicity such as fever that the researchers considered not to pose a safety risk to the subjects).

17. Have a history of immune deficiency, including a positive test for the human immunodeficiency virus (HIV), or suffer from other acquired or congenital immune deficiency diseases, or have a history of organ transplantation; 18. Active HBV or HCV infection or co-infection: If HBsAg (+) and/or HBcAb (+), HBV-DNA testing is required. The result must be less than 500 IU/mL or less than 2500 copies/mL or less than the upper limit of normal (ULN) for enrollment. For eligible subjects, if HBV-DNA can be detected, it is recommended that they receive nucleoside anti-hepatitis B virus treatment. If the HCV antibody is (+), HCV-RNA must be tested, and the result must be less than the upper limit of normal value (ULN) for enrollment. Subjects with co-infection of hepatitis B and C should be excluded (with positive HBsAg or HBcAb tests and positive HCV antibody tests).

19. Have received a live vaccine within 28 days prior to the first administration; 20. Pregnant or lactating women; 21. The researcher believes that the subjects have any clinical or laboratory test abnormalities or other reasons that make them unsuitable to participate in this clinical study.

22. Suffering from local or systemic diseases not caused by malignant diseases; Or diseases or symptoms caused by tumors that may lead to higher medical risks and/or uncertain survival assessment results, such as neoplastic leukemia-like reactions (white blood cell count > 20×109/L), cachexia manifestations (for example, known weight loss of more than 10% within 3 months before screening), etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
The Dose-Limiting Toxicity (DLT) of HLX37 within 21 days after the first Administration | From first dose to the end of Cycle 1 (each cycle is 3 weeks)
  DLT refers to the AEs that are determined to be related to the investigational product by the investigator, whose severity will affect the escalation of dose level. In this study, the DLT observation period lasts for 21 days after the first administration of HLX43.
2. The maximum tolerated dose (MTD) of HLX43 | From first dose to the end of Cycle 1 (each cycle is 3 weeks)
  The highest dose level, at which DLT is observed in no more than one of 6 evaluable patients, is defined as MTD of HLX43

SECONDARY OUTCOMES:
Objective response rate (ORR) | approximately up to 24 months
  Percentage of participants with complete response (CR) and partial response (PR) based on investigator assessment.
Duration of response (DOR) | approximately up to 24 months.
  Length of time response continued based on investigator's assessment.
Progression-free survival (PFS) | approximately up to 24 months.
  The PFS is defined as the time from the date of enrollment to the date of the first objective documentation of disease progression (as per RECIST v1.1) or death due to any cause,whichever occurred first.
Overall survival (OS) | approximately up to 24 months
  Time from the date of enrollment to the date of death for any cause.
Cmax | Up to 21 days after the first dose
  Maximum serum concentration (Cmax) of HLX37

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Chest Hospital, Shanghai
  - The Second Affiliated Hospital of Air Force Medical University of the People's Liberation Army of China, Xi'an

IPD SHARING:
Plan to Share IPD: No